CLINICAL TRIAL: NCT02749760
Title: The Effect of Dynamic Stabilizers for Valgus Stability of the Elbow in Professional Baseball Players
Brief Title: Prevention of Ulnar Collateral Ligament (UCL) Injuries in Minor League Pitchers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Bruce Toby, MD, Professor and Chair, Dept of Orthopedic Surgery and Sports Medicine, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY00000174
Record Dates: First submitted 2016-04-11; First posted 2016-04-25 (Estimated); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Elbow Injuries; Sprain Ulnar Collateral Ligament; Upper Extremity Injuries; Strain of Ulnar Collateral Ligament; Complete Tear Ulnar Collateral Ligament
Keywords: Ulnar collateral ligament; elbow injuries; dynamic elbow stabilizers; Tommy John's procedure; elbow injuries in pitchers
MeSH Terms: conditions — Elbow Injuries | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Minor league pitchers (Other): Minor league pitchers from a single professional baseball organization. Strength tests of the elbows will be administered at spring training and end of season for 5 years. If strength correlates to injury, strengthening and exercise programs may be established to target the stabilizers of the elbows.
  Interventions: Other: Strengthening program; Other: Exercise program

INTERVENTIONS:
Other: Strengthening program — Strengthening programs may be established to target the stabilizers of the elbows
Other: Exercise program — Exercise program may be established to target the stabilizers of the elbows.

SUMMARY:
This is a study of the muscle stabilizers of the elbow with respect to the prevention of Ulnar Collateral Ligament (UCL) injuries in pitchers. Pitchers are assessed at spring training and end of season for approximately 5 years. Pronator, flexor digitoum superficialis (FDS), and wrist flexion strength will be measured and correlated with upper extremity injuries and time missed from pitching. The investigators will also be measuring loss of strength over the season. The goal is to learn whether strength in these muscles prevents UCL injuries and finally whether these muscles can be strengthened to avoid such injuries.

DETAILED DESCRIPTION:
The goal of this study is to assess whether the strengths of the secondary muscular stabilizers toward valgus stress at the elbow, the wrist flexors, flexor digitorum superficialis, and pronator teres emanating from the medial epicondyle, affect the incidence of ulnar collateral ligament injuries of the elbows in pitchers. Pitchers in the minor leagues of a single professional baseball club will have the strength of these secondary muscular stabilizers assessed and then correlated to ulnar collateral ligament injuries and time missed from baseball season and subsequent seasons. A secondary goal is to assess whether strengthening exercises targeted toward these muscular stabilizers of the elbow can decrease the incidence of ulnar collateral ligament injuries in young baseball pitchers. This could impact the field by changing the emphasis from reconstruction and rehabilitation of ulnar collateral ligament injuries to prevention.

ELIGIBILITY:
Inclusion Criteria:

* Pitchers that are currently on a minor league baseball team.

Exclusion Criteria:

* Pitchers that currently have upper extremity injuries or are in active rehab for upper extremity injury.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2014-02; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
The Correlation of Strength to UCL Injuries in Minor League Pitchers | 5 years
  After measuring strength of elbow stabilizers for up to five years, we will determine whether strength correlates with UCL injuries.

SECONDARY OUTCOMES:
The Diminution of Strength in Minor League Pitchers | 5 years
  We will measure the diminution of strength over the course of a baseball season.

CONTACTS AND LOCATIONS:
Overall Officials: E B Toby, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anz AW, Bushnell BD, Griffin LP, Noonan TJ, Torry MR, Hawkins RJ. Correlation of torque and elbow injury in professional baseball pitchers. Am J Sports Med. 2010 Jul;38(7):1368-74. doi: 10.1177/0363546510363402. Epub 2010 Apr 16. PMID 20400752
- [Background] Azar FM, Andrews JR, Wilk KE, Groh D. Operative treatment of ulnar collateral ligament injuries of the elbow in athletes. Am J Sports Med. 2000 Jan-Feb;28(1):16-23. doi: 10.1177/03635465000280011401. PMID 10653538
- [Background] Bruce JR, Andrews JR. Ulnar collateral ligament injuries in the throwing athlete. J Am Acad Orthop Surg. 2014 May;22(5):315-25. doi: 10.5435/JAAOS-22-05-315. PMID 24788447
- [Background] Bruce JR, Hess R, Joyner P, Andrews JR. How much valgus instability can be expected with ulnar collateral ligament (UCL) injuries? A review of 273 baseball players with UCL injuries. J Shoulder Elbow Surg. 2014 Oct;23(10):1521-6. doi: 10.1016/j.jse.2014.05.015. PMID 25220199
- [Background] Conte SA, Fleisig GS, Dines JS, Wilk KE, Aune KT, Patterson-Flynn N, ElAttrache N. Prevalence of Ulnar Collateral Ligament Surgery in Professional Baseball Players. Am J Sports Med. 2015 Jul;43(7):1764-9. doi: 10.1177/0363546515580792. Epub 2015 Apr 29. PMID 25925603
- [Background] Costantino C, Vaienti E, Pogliacomi F. Evaluation of the peak torque, total work, average power of flexor-estensor and prono-supinator muscles of the elbow in baseball players. Acta Biomed. 2003 Aug;74(2):88-92. PMID 14509917
- [Background] Davidson PA, Pink M, Perry J, Jobe FW. Functional anatomy of the flexor pronator muscle group in relation to the medial collateral ligament of the elbow. Am J Sports Med. 1995 Mar-Apr;23(2):245-50. doi: 10.1177/036354659502300220. PMID 7778713
- [Background] Dugas JR, Ostrander RV, Cain EL, Kingsley D, Andrews JR. Anatomy of the anterior bundle of the ulnar collateral ligament. J Shoulder Elbow Surg. 2007 Sep-Oct;16(5):657-60. doi: 10.1016/j.jse.2006.11.009. Epub 2007 Jun 20. PMID 17583541
- [Background] Erickson BJ, Chalmers PN, Bush-Joseph CA, Verma NN, Romeo AA. Ulnar Collateral Ligament Reconstruction of the Elbow: A Systematic Review of the Literature. Orthop J Sports Med. 2015 Dec 9;3(12):2325967115618914. doi: 10.1177/2325967115618914. eCollection 2015 Dec. PMID 26740956
- [Background] Erickson BJ, Gupta AK, Harris JD, Bush-Joseph C, Bach BR, Abrams GD, San Juan AM, Cole BJ, Romeo AA. Rate of return to pitching and performance after Tommy John surgery in Major League Baseball pitchers. Am J Sports Med. 2014 Mar;42(3):536-43. doi: 10.1177/0363546513510890. Epub 2013 Dec 18. PMID 24352622
- [Background] Erickson BJ, Nwachukwu BU, Rosas S, Schairer WW, McCormick FM, Bach BR Jr, Bush-Joseph CA, Romeo AA. Trends in Medial Ulnar Collateral Ligament Reconstruction in the United States: A Retrospective Review of a Large Private-Payer Database From 2007 to 2011. Am J Sports Med. 2015 Jul;43(7):1770-4. doi: 10.1177/0363546515580304. PMID 26129959
- [Background] Fleisig GS, Andrews JR, Dillman CJ, Escamilla RF. Kinetics of baseball pitching with implications about injury mechanisms. Am J Sports Med. 1995 Mar-Apr;23(2):233-9. doi: 10.1177/036354659502300218. PMID 7778711
- [Background] Hamilton CD, Glousman RE, Jobe FW, Brault J, Pink M, Perry J. Dynamic stability of the elbow: electromyographic analysis of the flexor pronator group and the extensor group in pitchers with valgus instability. J Shoulder Elbow Surg. 1996 Sep-Oct;5(5):347-54. doi: 10.1016/s1058-2746(96)80065-6. PMID 8933456
- [Background] Haugstvedt JR, Berger RA, Berglund LJ. A mechanical study of the moment-forces of the supinators and pronators of the forearm. Acta Orthop Scand. 2001 Dec;72(6):629-34. doi: 10.1080/000164701317269076. PMID 11817880
- [Background] Jones KJ, Dines JS, Rebolledo BJ, Weeks KD, Williams RJ, Dines DM, Altchek DW. Operative management of ulnar collateral ligament insufficiency in adolescent athletes. Am J Sports Med. 2014 Jan;42(1):117-21. doi: 10.1177/0363546513507695. Epub 2013 Oct 21. PMID 24145949
- [Background] Keller RA, Steffes MJ, Zhuo D, Bey MJ, Moutzouros V. The effects of medial ulnar collateral ligament reconstruction on Major League pitching performance. J Shoulder Elbow Surg. 2014 Nov;23(11):1591-8. doi: 10.1016/j.jse.2014.06.033. Epub 2014 Aug 31. PMID 25183663
- [Background] Laudner KG, Wilson JT, Meister K. Elbow isokinetic strength characteristics among collegiate baseball players. Phys Ther Sport. 2012 May;13(2):97-100. doi: 10.1016/j.ptsp.2011.06.007. Epub 2011 Aug 24. PMID 22498150
- [Background] Lin F, Kohli N, Perlmutter S, Lim D, Nuber GW, Makhsous M. Muscle contribution to elbow joint valgus stability. J Shoulder Elbow Surg. 2007 Nov-Dec;16(6):795-802. doi: 10.1016/j.jse.2007.03.024. Epub 2007 Nov 1. PMID 17936028
- [Background] Park MC, Ahmad CS. Dynamic contributions of the flexor-pronator mass to elbow valgus stability. J Bone Joint Surg Am. 2004 Oct;86(10):2268-74. doi: 10.2106/00004623-200410000-00020. PMID 15466738
- [Background] Morrey BF, Tanaka S, An KN. Valgus stability of the elbow. A definition of primary and secondary constraints. Clin Orthop Relat Res. 1991 Apr;(265):187-95. PMID 2009657
- [Background] Otoshi K, Kikuchi S, Shishido H, Konno S. The proximal origins of the flexor-pronator muscles and their role in the dynamic stabilization of the elbow joint: an anatomical study. Surg Radiol Anat. 2014 Apr;36(3):289-94. doi: 10.1007/s00276-013-1168-3. Epub 2013 Jul 25. PMID 23884470
- [Background] Udall JH, Fitzpatrick MJ, McGarry MH, Leba TB, Lee TQ. Effects of flexor-pronator muscle loading on valgus stability of the elbow with an intact, stretched, and resected medial ulnar collateral ligament. J Shoulder Elbow Surg. 2009 Sep-Oct;18(5):773-8. doi: 10.1016/j.jse.2009.03.008. Epub 2009 May 31. PMID 19487136
- [Background] Werner SL, Fleisig GS, Dillman CJ, Andrews JR. Biomechanics of the elbow during baseball pitching. J Orthop Sports Phys Ther. 1993 Jun;17(6):274-8. doi: 10.2519/jospt.1993.17.6.274. PMID 8343786